CLINICAL TRIAL: NCT06165783
Title: The Effect of Therapeutic Exercises and Ultrasound for Rehabilitation of Partially Injured Hamstring Muscles in Elite Football Players: a Study Protocol for a Randomized Controlled Trial
Brief Title: Rehabilitation of Partially Injured Hamstring Muscles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Kamal Hadib Abdulridha, Principal Investigator, Universidad de Zaragoza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Injured Hamstring Muscles
Record Dates: First submitted 2023-11-23; First posted 2023-12-11 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Hamstring Injury
Keywords: Therapeutic exercises, Hamstring muscle injuries, TUS; Therapeutic exercises; Hamstring muscle injuries; TUS
MeSH Terms: interventions — Exercise Therapy; High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- evaluate the effect of using therapeutic exercises and ultrasound (Experimental): evaluate the effect of using therapeutic exercises and ultrasound for the rehabilitation of partially injured hamstring muscles.
  Interventions: Other: Therapeutic Exercises and Ultrasound
- analyse its effectiveness on the speedy healing (Experimental): analyse its effectiveness on the speedy healing, which will be defined through some physical variables (hamstring muscle strength, the electrical activity of hamstring muscles) and pain perception.
  Interventions: Other: Therapeutic Exercises and Ultrasound

INTERVENTIONS:
Other: Therapeutic Exercises and Ultrasound — describe the rationale and methodology for evaluating the effect of using therapeutic exercises and ultrasound in the rehabilitation of partially injured hamstring muscles

SUMMARY:
The aim of this study protocol is to describe the rationale and methodology for evaluating the effect of using therapeutic exercises and ultrasound in the rehabilitation of partially injured hamstring muscles on elite football players.

DETAILED DESCRIPTION:
Hamstring muscle injuries are common among highly active individuals. Modern Football is a challenging sport characterized by extremely dynamic and cyclical game motions including numerous bouts of high-speed movements such as accelerating, jumping, and change in direction, all of which are carried out at a high level of physical and technical difficulty. The most common reason for hamstring muscle injury is high-performance intensity. In addition, neuromuscular fatigue, athlete aging, low muscle strength, and hamstring muscle flexibility are also risk factors for hamstring muscle injuries. On the other hand, the main causes of repetition injury to the same muscle are the presence of a previous injury, the size of the muscle tear and the lessening of the long head muscle bundles of the biceps femoris

ELIGIBILITY:
Inclusion criteria:

* Players from the eight clubs in the Iraqi Football League
* Partially strained hamstring muscle pain when training football or playing a match, identified as:

  a. Player reported sudden pain in hamstring muscle c. Without any additional ailment.
* Based on the clinical signs and symptoms, defined as:

  1. Localised pain when palpating of hamstring muscle
  2. Localised pain from at least one of the following activities: The Extender, The Diver, and The Glider.
* MRI-confirmed of partially injured hamstring
* Available for follow-up

Exclusion criteria:

* Players with other injuries apart from hamstring injuries
* Players with a recent six-month history of a verified or suspected hamstring injury in the same leg.
* injured players who are already taking part in another rehabilitation program
* General contraindications for MRI

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Male
Enrollment: 24 (Actual)
Dates: Start 2024-03-21 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Time to return to play | Daily session from first therapy session until moment of return to play, up to an average of Six Weeks
  The primary outcomes will be speedy healing, that is, the amount of time needed to recover from an injury in order to fully participate in team training and be available for match selection by the medical staff based on five standardized criteria: 1. no pain on palpation 2. pain free Range of Motion (ROM) 3. Muscular strength evaluation 4. Symptom-free completion of rehabilitation program 5. A specific running test.

SECONDARY OUTCOMES:
Hamstring muscle strength | Daily session from first therapy session until moment of return to play, up to an average of Six Weeks
  Force Sensor from Chronojump. Is an sensor measure of to conduct isometric knee flexion strength testing at two distinct angles: 15° and 90° of knee flexion.
Muscle bio potential signals | Daily session from first therapy session until moment of return to play, up to an average of Six Weeks
  The Electromyogram (EMG) is collected at 1000 Hz with MyoTrace™ 400 . Is a versatile portable handheld, Self-adhesive silver chloride dual snap electrodes for surface attachment will be placed on the leg muscles. The MyoTrace 400 handheld transmitter.
Degree of pain | Daily session from first therapy session until moment of return to play, up to an average of Six Weeks
  Pain visual analog scale (VAS). It is a unidimensional measure of hamstrings pain intensity that consists of a straight horizontal line of fixed length (typically 100 mm) that is graduated. The ends, which were towards the direction of left (worse) to right (best), defined the extreme boundaries of the parameter to be calculated (pain); the higher the score, the more severe the suffering.

CONTACTS AND LOCATIONS:
Overall Officials: Kamal H Abdulridha, PhD/Studet, Principal Investigator — Universidad de Zaragoza
Locations (1):
- University of Baghdad/ college of Physical Education and Sports Sciences, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No